CLINICAL TRIAL: NCT04037410
Title: Effects of Environmental Temperature on White Adipose Tissue Thermogenic Capacity of Cancer Patients
Brief Title: Environmental Temperature and White Adipose Tissue in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Petros Dinas (Other)
Responsible Party: Sponsor-Investigator, Petros Dinas, Senior Researcher in human physiology, University of Thessaly
Organization: University of Thessaly (Other)
Other Study IDs: 2. Tenv & cancer patient
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Cancer Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to retrospectively identify the association between the thermogenic capacity of white adipocytes and the environmental temperature, in cancer patients.

DETAILED DESCRIPTION:
Obesity is characterized by excessive white adipose tissue (WAT) that increases risk for disease. About 700 million adults are obese worldwide, designating the need of reducing excessive WAT in humans and subsequently the risk for disease. For this reason, previous research focused on the thermogenic capacity of white adipocytes in response to cold exposure. Cold exposure represents a main stimulus for increased thermogenic capacity in human white adipocytes, which may have an impact on body weight loss and subsequently on obesity phenomenon.

In a cohort of 202 cancer patients (male=126), who undertook a Positron Emission Tomography (PET/CT), we retrospectively investigated the association between Tenv and thermogenic capacity of subcutaneous WAT (dorsolumbar region near vertebrae L3 and abdominal region). These patients undertook a PET/CT examination in order to define their disease status. They were given instructions in advance to refrain from smoking, exercise and excessive muscle stressors 24-hour prior to their examination. On the day of the measurements they advised to transport themselves by car to the PET/CT Laboratory between 08:00 am to 12 pm, following at least a 6-hour fasting. Patients were first injected an appropriate dose of 18F-FDG (based on their body weight) and then they were remained in a sitting relaxed position within a quiet room of 22-24°C for 60 minutes. Following this period, patients undertook the PET/CT examination, which included on average eight bed positions, while four minutes scanning per bed position was used.

PET/CT imaging analysis for WAT activity (dorsolumbar region near vertebrae L3 and abdominal region) was performed by two independent trained physicians, using previous methodology.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients who undertook a PET/CT examination independently of their disease status

Exclusion Criteria:

* Examinations prior to 2016

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients independently of their disease status
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Assessment of thermogenic capacity of white adipocytes | The SUV of white adipocytes for each patient was measured once via the PET/CT software between 10-30 May 2019.
  Thermogenic capacity of white adipocytes was measured via Positron Emission Tomography/computed tomography (PET/CT) device, unit of measurement: Standardized Uptake Value (SUV)
Environmental temperature | The daily environmental temperature was obtained from Weather Underground (www.wunderground.com) on the 10th May 2019
  The daily environmental temperature was obtained in degrees Celsius for the period 1-1-2016 to 30-4-2019.

CONTACTS AND LOCATIONS:
Locations (1):
- Petros Dinas, Trikala, Thessaly, Greece